CLINICAL TRIAL: NCT07017049
Title: Effects of Integrative Neuromuscular Traning on Physical Fitness and Dribbling Performance Among High School Male Football Players in Shandong, China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinrui Zhang (Other)
Responsible Party: Sponsor-Investigator, Xinrui Zhang, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024065
Record Dates: First submitted 2025-04-30; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Adolescent; Healthy Volunteers (HV); Physical Fitness and Technical Skills; Football Players
Keywords: integrative neuromuscular training; football players; adolescent; physical fitness; drilling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- integrative neuromuscular training (Experimental): Participants in this arm will complete a 12-week integrative neuromuscular training (INT) program, 3 times per week, 1 hour per session. The program includes progressive balance, strength, plyometric, speed, agility, and coordination exercises. Weeks 1-2 focus on threshold training (55-65% HRmax), including single-leg balance, box jumps (30 cm), squats, and sprints. Weeks 3-5 increase intensity (65-75% HRmax) with BOSU balance, loaded jumps, lunges, and agility drills. Weeks 6-8 and 9-12 emphasize high-threshold training (70-85% HRmax), with BOSU dynamic balance, 50 cm jumps, triangle and square jumps, Bulgarian squats, sprints, and shuttle runs with ball handling. Rest: 30-60 sec between sets.
  Interventions: Behavioral: Integrative Neuromuscular Training
- Routine training intervention (Active Comparator): Participants in the control group will follow the standard physical training program of the school over a 12-week period, with sessions conducted 3 times per week, each lasting approximately 50 minutes (including warm-up and cool-down). The training intensity will progressively increase from 55%-65% HRmax in weeks 1-3, 65%-75% HRmax in weeks 4-8, and 75%-85% HRmax in weeks 9-12.
  Each session includes:
  Warm-up (10 minutes): Movement of hands and legs, small-sided games, ball handling, and stretching exercises.
  Intervention (30 minutes):
  Weeks 1-3: Barbell back squat, barbell deadlift, bench press, continuous broad jumps, continuous burpee jumps, frontal plank (60 sec), 50m sprinting (5 reps), 2 sets of each exercise with 30-60 seconds rest.
  Weeks 4-5: Similar structure with increased repetitions (barbell exercises 6-10 reps, plank 70 sec).
  Weeks 6-8: Barbell back squat, deadlift, bench press, broad jumps, each for 3 sets, 30-60 sec rest.
  Weeks 9-12: Higher load with 8-12 reps pe
  Interventions: Behavioral: Routine training intervention

INTERVENTIONS:
Behavioral: Integrative Neuromuscular Training — Participants will receive a 12-week Integrative Neuromuscular Training (INT) program, conducted 3 times per week, each session lasting 1 hour. The intervention includes progressive exercises targeting balance, strength, plyometrics, speed, agility, and coordination. Training intensity increases from 55-65% HRmax in weeks 1-2, to 65-75% HRmax in weeks 3-5, and 70-85% HRmax in weeks 6-12. Exercises include single-leg balance, BOSU balance, box jumps (30-50 cm), lateral jumps, squats, Nordic hamstring exercises, sprints (20-30m), shuttle runs, and agility drills. Rest between sets is 30-60 seconds.
  Arms: integrative neuromuscular training
Behavioral: Routine training intervention — Participants in the control group will follow the standard physical training program of the school over a 12-week period, with sessions conducted 3 times per week, each lasting approximately 50 minutes (including warm-up and cool-down). The training intensity will progressively increase from 55%-65% HRmax in weeks 1-3, 65%-75% HRmax in weeks 4-8, and 75%-85% HRmax in weeks 9-12.
  Each session includes:
  Warm-up (10 minutes): Movement of hands and legs, small-sided games, ball handling, and stretching exercises.
  Intervention (30 minutes):
  Weeks 1-3: Barbell back squat, barbell deadlift, bench press, continuous broad jumps, continuous burpee jumps, frontal plank (60 sec), 50m sprinting (5 reps), 2 sets of each exercise with 30-60 seconds rest.
  Weeks 4-5: Similar structure with increased repetitions (barbell exercises 6-10 reps, plank 70 sec).
  Weeks 6-8: Barbell back squat, deadlift, bench press, broad jumps, each for 3 sets, 30-60 sec rest.
  Weeks 9-12: Higher load with 8-12 reps per
  Arms: Routine training intervention

SUMMARY:
This study investigates the effects of a 12-week Integrative Neuromuscular Training (INT) program on physical fitness, balance, and dribbling skills in male high school soccer players in Shandong, China. INT, which combines strength, agility, balance, core stability, and proprioception, has been shown internationally to enhance athletic performance and prevent injuries among youth athletes. While widely applied in sports like basketball, volleyball, and swimming abroad, research on INT in Chinese male soccer players remains limited.

A total of 60 male soccer players (aged 16-18) with at least two years of training experience will be recruited from two high schools in Jinan and divided equally into experimental and control groups. The experimental group will undergo INT three times per week for 12 weeks, while the control group will continue regular soccer training. The study will measure changes in strength, speed, endurance, flexibility, static and dynamic balance, and dribbling performance. Data collection spans 16 weeks, including pre-tests, intervention, and post-tests. Statistical analysis will be conducted using SPSS 26.0, employing descriptive statistics, GEE models, and repeated measures ANOVA. This research aims to provide scientific evidence for the use of INT in youth soccer training in China.

DETAILED DESCRIPTION:
Integrative Neuromuscular Training (INT) is a comprehensive and multi-faceted training model that integrates strength, agility, balance, core stability, and proprioception. In recent years, the application of INT has gained increasing attention among youth athletes due to its effectiveness in enhancing physical fitness and athletic performance. Studies have shown that INT not only improves fitness parameters but also plays a significant role in injury prevention.

International research has demonstrated the widespread use of INT in sports such as basketball, volleyball, and swimming. These studies highlight that INT significantly enhances lower limb strength, dynamic balance, speed, and agility.

However, in China, particularly among high school male soccer players, research on INT remains limited. This study aims to fill this gap by exploring the effects of a 12-week INT program on physical fitness (including strength, speed, endurance, and flexibility), balance (both static and dynamic), and dribbling skills in high school male soccer players in Shandong Province. The objective is to provide scientific evidence and empirical data to support the integration of INT into youth soccer training programs in China.

The study will recruit 60 male high school soccer players, aged 16-18, from two high schools in Jinan, Shandong. Participants must have at least two years of soccer training experience and be in good health, with no chronic conditions or injuries affecting performance. Those with a history of severe sports injuries or currently undergoing rehabilitation or medical treatment will be excluded. The participants will be randomly assigned to either an experimental group or a control group, with 30 players in each.

The research will span approximately 16 weeks. The first two weeks will involve pre-testing, equipment calibration, and baseline measurements. Weeks 3 to 14 will be the intervention period, during which the experimental group will undergo INT three times per week, while the control group will continue with their regular soccer training. In the final two weeks, post-tests and data analysis will be conducted.

Physical fitness will be assessed through tests such as squat strength, standing long jump, Yo-Yo endurance test, 10m and 20m sprints, Illinois agility test, and sit-and-reach flexibility. Balance will be evaluated using the Y-Balance test and single-leg eyes-closed stance. Soccer-specific skills will be measured using 20m straight-line dribbling and zig-zag dribbling tests. Data will be analyzed using SPSS 26.0, including descriptive statistics (mean ± standard deviation), between-group comparisons using Generalized Estimating Equations (GEE), and repeated measures ANOVA to assess changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Male high school football players aged between 16 to 18 years
2. Regular participation in football training without prior structured neuromuscular warm-up training experience within the last 12 months
3. Physically healthy and capable of performing all required tests
4. Voluntary consent to participate in all assessments and training sessions
5. Clear understanding of the objectives and procedures of the study

Exclusion Criteria:

1. History of significant musculoskeletal injuries (e.g., knee, ankle, or hip injuries) within the previous year
2. Presence of current health conditions or medication use that might interfere with physical performance or muscular activity
3. Any neurological disorders or chronic health issues that could impact participation in training or assessment
4. Previous experience with structured neuromuscular warm-up training within the last year
5. Uncertainty regarding the ability to consistently attend and complete the training due to personal or external factors

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Physical fitness (Sprint Speed) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Sprint speed was measured as the time (in seconds) to complete a 10-meter sprint from a standing start on a standard track, using a digital stopwatch.
  The best time from two attempts was recorded.
Physical fitness (muscle strength) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Lower limb muscle strength was measured by the maximum load lifted in a back squat using a standard barbell and weight plates. The results are reported in kilograms (kg), with participants performing up to their one-repetition maximum (1RM).
Physical fitness (explosive power) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Explosive power was measured by the height of a countermovement jump (CMJ) using a jump mat or force platform. The highest jump from two attempts was recorded in centimeters (cm).
Physical fitness (Agility) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Agility was assessed by timing how long participants took to complete the Illinois Agility Test course, measured in seconds. The test was conducted on a standard layout with electronic timing gates.
Physical fitness (Flexibility) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Flexibility was measured by the Sit-and-Reach Test using a standard sit-and-reach box. The maximum reach distance was recorded in centimeters (cm), with the best of two attempts used for analysis.
Dribbling performance in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Dribbling agility was measured using the Illinois Agility Test while dribbling a football. Time to complete the course was recorded in seconds using electronic timing gates.
Anthropometric (height) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Height was measured using a standard stadiometer, with results given in centimeters (cm) accurate to 0.1 cm. Participants stood barefoot with heels together for the measurement.
Anthropometric (weight) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Weight was measured using a calibrated electronic scale, with results given in kilograms (kg) accurate to 0.1 kg. Participants wore light clothing and no shoes.
Anthropometric (Body Mass Index) in high school football players | baseline, after 6 weeks of intervention, and post-intervention at week 12
  Body Mass Index (BMI) was calculated as weight in kilograms divided by the square of height in meters (kg/m²). Weight was measured using a digital scale (accurate to 0.1 kg), and height was measured with a stadiometer (accurate to 0.1 cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Jigang Senior High School，46 Sangyuan Rd, Licheng District, Jinan, Jinan, Shandong, China, 250100, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to privacy concerns and ethical considerations, as the participants are minors. Data sharing may pose a risk to participant confidentiality, and there is no consent obtained for public data sharing.

REFERENCES:
- [Background] Xiong J, Li S, Cao A, Qian L, Peng B, Xiao D. Effects of integrative neuromuscular training intervention on physical performance in elite female table tennis players: A randomized controlled trial. PLoS One. 2022 Jan 20;17(1):e0262775. doi: 10.1371/journal.pone.0262775. eCollection 2022. PMID 35051233
- [Background] Hammami R, Negra Y, Nebigh A, Ramirez-Campillo R, Moran J, Chaabene H. Preseason Integrative Neuromuscular Training Improves Selected Measures of Physical Fitness in Highly Trained, Youth, Male Soccer Players. J Strength Cond Res. 2023 Jun 1;37(6):e384-e390. doi: 10.1519/JSC.0000000000004394. Epub 2022 Nov 30. PMID 37235541